CLINICAL TRIAL: NCT06422728
Title: The Effectiveness of Transdiagnostic CBT Protocol on Anxiety Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Haldun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-71395021-050.06.04-35012
Record Dates: First submitted 2024-05-14; First posted 2024-05-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anxiety Disorders; Social Anxiety Disorder; Generalized Anxiety Disorder; Panic Disorder; Anxiety Disorder NOS
Keywords: transdiagnostic approach; unified protocol,; anxiety disorders; CBT; cognitive behavioral therapy
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Generalized Anxiety Disorder; Panic Disorder

STUDY DESIGN:
Intervention Model Description: This study will search the effectiveness of the unified protocol on anxiety disorders. For this purpose, there will be an intervention group (unified protocol will be applied) and a control group. The participants will be assigned randomly to the groups.
Who Masked: Participant
Masking Description: In this study, single-blind procedure will be applied to reduce biases. For this purpose, participants will be informed only about the general procedure of group therapy (e.g. general focus of the group therapy, number of sessions, duration of sessions, number of participants) but will not be informed about which intervention they receive and which group they are assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdiagnostic Unified Protocol (Experimental): The intervention group will receive the transdiagnostic unified protocol (UP) for anxiety disorders that is developed in this study. The UP is based on CBT model and will last for 8 weeks and there will be a follow-up session after one month. Each session will last 1 and a half hours. The pre-, post- and follow-up tests will be given to them to test the effectiveness of the UP.
  Interventions: Other: Unified Protocol for Anxiety Disorders
- Client-Centered Supportive Therapy (Active Comparator): The supportive therapy group will also last for 8 weeks and there will be a follow-up session after one month. Each session will last 1 and a half hours. The pre-, post- and follow-up tests will be given to them, too.
  Interventions: Other: Client-centered Supportive Therapy

INTERVENTIONS:
Other: Unified Protocol for Anxiety Disorders — The UP is planned in group therapy format and includes interventions on common transdiagnostic features. The sessions in the protocol are planned as follows:
  Session 1 - Assessment: introduction, talking on group rules and the process, setting goals
  Session 2 - Psychoeducation: the CBT model is introduced.
  Session 3 - Emotions: the role of emotions are discussed.
  Session 4, 5 & 6 - Thoughts: the role of thoughts is mentioned. The participants learn to challenge unfunctional thoughts and generate alternative explanations. Also, exercises on excessive worry are applied.
  Session 7 - Behaviors: the role of behaviors and the things that can/cannot be controlled are discussed.
  Session 8 - Evaluation & Maintaining Accomplishments: includes a review of what has been learnt during the group therapy and an evaluation on maintaining the accomplishments.
  Session 9 - Follow-up session: one month later.
  Arms: Transdiagnostic Unified Protocol
Other: Client-centered Supportive Therapy — Client-entered therapy provides a non-directive supportive environment for the participants, that includes reflective listening and nonjudgmental and empathic communication. In this group, no CBT intervention will be applied. Through the supportive and non-directive environment, only the effect of relationship will be investigated as a common factor in psychotherapy.
  Arms: Client-Centered Supportive Therapy

SUMMARY:
The transdiagnostic approach argues that the common features are needed to be taken into account [e.g. distress intolerance (DI), intolerance of uncertainty (IU), worry)] underlying emotional disorders rather than evaluating them separately due to the fact that the dissection of anxiety disorders has increased with each emerging version of the Diagnostic and Statistical Manual of Mental Disorders (DSM), in which the classification of anxiety disorders resulted in an increased number of intervention protocols for each disorder. This also caused an increase of comorbidity among anxiety disorders. Transdiagnostic approach offers a unified protocol (UP) for strengthening the common features, and thereby both preventing the emergence of emotional disorders or intervening the symptom severity of emotional disorders, which can be applied to different types of emotional disorders. The main aim of this study is to develop a UP which is planned to be applied as a group therapy. The UP will include interventions developing the levels of common transdiagnostic features (DI, IU and worry). The study's second aim is to investigate the effect of the developed UP on DI, IU and worry. The third one is to search the effect of the developed UP on symptom severity levels of anxiety disorders. Fourthly, this study will search if the levels of transdiagnostic common features (DI, IU and worry) will predict the levels of symptom severity of anxiety disorders'.

DETAILED DESCRIPTION:
The transdiagnostic approach argues that common features are needed to be taken into account [e.g. distress intolerance (DI), intolerance of uncertainty (IU), worry] underlying emotional disorders rather than evaluating them separately since the dissection of anxiety disorders has increased with each emerging version of the Diagnostic and Statistical Manual of Mental Disorders (DSM), in which the classification of anxiety disorders resulted in an increased number of intervention protocols for each disorder. That is why an increase in comorbidity among anxiety disorders is observed. The transdiagnostic approach offers a unified protocol (UP) for strengthening the common features, thereby preventing the emergence and intervening in several emotional disorders.

As part of dissertation, the main aim of this study is to develop UP in Turkish, and measure the effectiveness of the UP on anxiety disorders and the transdiagnostic features. The UP is planned in group therapy format and includes interventions strengthening the common transdiagnostic features (DI, IU, and worry). This protocol is based on cognitive behavioral therapy (CBT) model. The sessions in the protocol are planned as follows:

Session 1 is assessment session and Session 2 is on psychoeducation, which mainly intend to introduce the CBT model. In session 3, emotions are discussed, revealing that emotions point out what is important for us in life. In session 4, 5 and 6, thoughts are worked on. The participants learn to deal with worry and to challenge unfunctional thoughts and generate alternative explanations. Session 7 focuses on behaviors, in which the role of behaviors and the things that can/cannot be controlled are discussed. Session 8 includes a review of what has been learnt during the group therapy and an evaluation on maintaining the accomplishments. In addition, a follow-up session is planned after one month.

In this study, there will be an intervention (UP) group and a control group. The participants will be assigned to the groups randomly. The measurements are the Distress Intolerance Scale (DTS), Intolerance of Uncertainty Scale-12 (IUS-12), Penn State Worry Questionnaire (PSWQ), Metacognitions Questionnaire-30 (MCQ-30), Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder Assessment (GAD-7).

The uniqueness of this protocol is to be the first UP in Turkish with its own order. It is expected to promote transdiagnostic studies in Turkey. This research is also important in contributing to the literature on transdiagnostic studies, which offer an alternative to comorbidity and a decrease in the symptom severity of anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with at least one of the following disorders in the pre-interview (SCID 5 interview for diagnosis): generalized anxiety disorder (GAD), panic disorder (PD), social anxiety disorder (SAD) or anxiety disorder not otherwise specified (NOS).

Exclusion Criteria:

* Active substance use or having a psychiatric history related to substance use
* Having a co-diagnosis of psychotic disorders or bipolar disorders
* Receiving active psychotherapy support
* Being not graduated from primary school

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | pre-test (baseline at Week 1), post-test (at Week 8), follow-up test (1 month after post-test)
  Generalized Anxiety Disorder-7 (GAD-7) scale will be used to measure anxiety level. GAD-7 is a self-report scale consisting of 7 items. It is a 4-point Likert type scale. Items are scored between 0 (Not at all) and 3 (Nearly every day). Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety. In the total score, the cut-off score for GAD diagnosis is 10.
Distress Tolerance | pre-test (baseline at Week 1), post-test (at Week 8), follow-up test (1 month after post-test)
  Distress Tolerance Scale (DTS) scale will be used to measure distress tolerance level. DTS consists of a total of 15 items. Each item is rated on a 5-point Likert scale range from 1 (Strongly disagree) to 5 (Strongly disagree). A low total score indicates low distress tolerance level.
Intolerance of Uncertainty | pre-test (baseline at Week 1), post-test (at Week 8), follow-up test (1 month after post-test)
  Intolerance of Uncertainty Scale (IUS) - Short Version will be used to measure the level of intolerance of uncertainty. IUS-12 is a self-report scale consisting of 12 items in total. It is a 5-point Likert scale. Each item is scored between 1 (not at all characteristic of me) to 5 (entirely characteristic of me). A high total score indicates a high level of intolerance to uncertainty.
Worry | pre-test (baseline at Week 1), post-test (at Week 8), follow-up test (1 month after post-test)
  Penn State Worry Questionnaire will be used to measure the level of worry. PSWQ is a self-report scale with a 5-point Likert-type, consisting of a total of 16 items. Scale items are scored between 1 (Not at all typical) - 5 (Very typical of me). An increase in the PSWQ total score indicates a high level of worry.
Metacognition | pre-test (baseline at Week 1), post-test (at Week 8), follow-up test (1 month after post-test)
  Metacognition Questionnaire-30 Short Form will be used to measure metacognitive beliefs. MCQ-30, consisting of a total of 30 items, has a 4-point Likert-type scale. Each item is scored between 1 (Do not agree) and 4 (Agree very much). An increase in scale scores indicates an increase in pathological metacognitive activity.
Depression | pre-test (baseline at Week 1), post-test (at Week 8), follow-up test (1 month after post-test)
  Patient Health Questionnaire-9 (PHQ-9) will be used to measure the level of depression. PHQ-9 consists of 9 questions which is a 4-point Likert type scale. Each item is scored between 0 (Not at all) - 3 (Nearly every day). As the total score increases, the severity of depression increases.

CONTACTS AND LOCATIONS:
Overall Officials: Iclal AYDIN, MA, Principal Investigator — İbn Haldun University
Locations (1):
- Iclal AYDIN, Zeyti̇nburnu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share because of the ethical concerns of the participants' privacy.